CLINICAL TRIAL: NCT05804266
Title: A Randomized Comparison of UnderwateR Versus Regular Coagulation in Endoscopic Submucosal DissectioN and Third Space Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CURRENT ID 3303
Record Dates: First submitted 2023-03-08; First posted 2023-04-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Diseases; Endoscopic Surgery
Keywords: POEM, TSE, G-POEM, Z-POEM, PREM
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Considering a mean number of treated vessel of 4 per each patient, with standard technique we expect that 36% of patients need will have at least on vessel bleeding and requiring an adjunctive hemostasis, versus 6% of patients with underwater coagulation technique. With an alpha error of 5%, a power of 80% we need a total of 70 patients (35 in each arm), to detect this difference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional coagulation of vessels (Active Comparator): during study procedure accomplished under CO2-insufflation with the HK using SWIFT COAG E3, 89 W for POEM and SWIFT COAG E4, 124 W for ESD
  Interventions: Procedure: Coventional coagulation
- Underwater coagulation of vessels (Experimental): during study procedure carried out in the underwater setting with the HK using SWIFT COAG E3, 89 W for POEM and SWIFT COAG E4, 124 W for ESD
  Interventions: Procedure: Underwater coagulation

INTERVENTIONS:
Procedure: Coventional coagulation — In the conventional group, the haemostasis of vessels will be performed with the conventional coagulation technique under CO2 insufflation. First, submucosal fibres surrounding a blood vessel will be dissected and the vessel will be isolated. After, both sides of the isolated vessel will be coagulated using SWIFT COAG E3, 89 W for POEM and SWIFT COAG E4, 124 W for ESD until the blood vessel turns white and can be finally cut.
  Arms: Conventional coagulation of vessels
Procedure: Underwater coagulation — In the treatment group, the prophylactic haemostasis of vessels will be accomplished by the underwater coagulation technique. First, physiological solution will be instilled until there is no more air around the blood vessel. Then, the vessel will be coagulated using SWIFT COAG E3, 89 W for POEM and SWIFT COAG E4, 124 W for ESD until it turns white and, after the removal of all the physiological solution, can be finally cut.
  Arms: Underwater coagulation of vessels

SUMMARY:
What the investigatorpropose in this protocol is a technique already used in clinical practice. It prevents the risk of bleeding and make third space endoscopy easier, quicker, safer and cheaper. Indeed, we noticed that preventive underwater coagulation of the candidate vessels during the submucosal dissection with the Hybrid Knife (HK), seal the wall of the vessel, resulting in a subsequent cut under CO2 without any bleeding. Such preventive coagulation is likely to be related with the conduction of the current underwater as it focalizes all the power on the interface between the vessel and the water, allowing a soft sealing of the vessel without cutting it. Despite widely used, there is no evidence up to know on the benefit and harm of such coagulation technique.

The hypothesis is that the use of this approach in clinical practice, especially when used to coagulate a vessel, may lead to an increase in safety, feasibility and cost-effectiveness, reducing the procedural time, the rate of complications and the need for coagulation forceps in comparison with the conventional preventive coagulation technique under CO2 insufflation. Therefore, this randomized study compares the underwater coagulation technique with the conventional coagulation technique in the CO2 setting during the submucosal dissection in third space endoscopy.

DETAILED DESCRIPTION:
POEM will be performed under general anaesthesia in the supine position. The location of the esophagogastric junction (EGJ) will be identified and, then, after submucosal injection of saline mixed with methylene blue, a 2-cm mucosal incision carried out at 5-6 o'clock position about 10 cm above the EGJ. After, a dissection of the underlying submucosa will be performed to access the submucosal space. Then, the dissection of the submucosal layer will be continued to create the submucosal tunnel down to the narrower submucosal space at the EGJ and 2-3 cm into the cardia. During the submucosal tunnelling, coagulation of vessels will be performed with HK using SWIFT COAG E3, 89 W in the underwater setting in the treatment arm or with the standard technique in the CO2-setting in the conventional group. After, the myotomy of the circular muscular layer will be performed from 2-3 cm below the mucosal incision until 2-3 cm below the EGJ in both groups. In some cases, a full thickness myotomy, including the longitudinal muscular layer, will be carried out. Finally, complete closure of the mucosal entry site will be achieved with haemostatic clips. The procedure time, the number of instrument exchanges and bleeding episodes requiring the use of coagulation forceps during the procedure will be documented from start of submucosal tunnelling until final clip closure in both groups.

Fujifilm high-definition gastroscopes (Fujifilm Co., Tokyo, Japan) with a 2.8-mm operative channel and a transparent distal cap attachment will be used in both groups. A submucosal lift with saline mixed with methylene blue through a 23 G injection needle will be accomplished for the mucosal entry. POEM will be carried out using a HK (Erbe Elektromedizin GmbH, Tübingen) in both groups. This instrument has an outer diameter of 2.1 mm and an inner diameter of 1.2 mm with both electrosurgical and water-jet (WJ) surgery technologies in one device. The HK combines needle-less submucosal injection, cutting, dissection and coagulation in one instrument. The modular VIO generator (VIO 3, Erbe Elektromedizin GmbH, Tübingen, Germany) will be used as an electrosurgical system in combination with the ERBEJet 2 WJ surgery system in both groups. A slightly methylene blue-stained isotonic saline solution will be used for submucosal injection with the WJ technique in both groups. Mucosal incision and myotomy will be carried out using ENDO CUT Q 2-3-3 and ENDO CUT Q 2-3-3, respectively, in both groups.

ELIGIBILITY:
Inclusion criteria:

All >18 years-old patients undergoing ESD for superificial GI neoplastic lesions or POEM for esophageal achalasia

Exclusion criteria:

patients on antithrombotic/anticoagulant therapy patients suffering from bleeding disorders patients with esophageal and/or gastric varices patients previously treated for the same reason patients who were not able or refused to give informed written consent. vessels smaller than the knife inner diameter (1.2 mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Bleeding | 12 months
  Rate of patients with at least on vessel bleeding and requiring an adjunctive hemostasis

SECONDARY OUTCOMES:
delayed bleeding | 12 months
  Rate of delayed bleeding per patient defined as clinical evidence of bleeding (hematemesis, hematochezia or melena or a decrease of hemoglobin concentration > 2g/dL) which required transfusion or endoscopic reintervention with hemostasis within 30 days of hospital discharge the endoscopic resection.
instrument exchanges | 12 months
  Number of instrument exchanges per procedure
complications rate | 12 months
  Other intra- and post-procedural complications rate per patient
Procedural time | 12 months
  Mean procedural time
Patient-reported outcomes | 12 months
  in terms of tolerability and post-procedural pain
variation of blood values | 12 months
  Mean percentage variation of haematocrit, haemoglobin, C-reactive protein and white blood cells
intra-procedural bleeding | 12 months
  Rate of intra-procedural bleeding per each vessel requiring the use of coagulation forceps

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inoue H, Navarro MJH, Shimamura Y, Tanabe M, Toshimori A. The Journey from Endoscopic Submucosal Dissection to Third Space Endoscopy. Gastrointest Endosc Clin N Am. 2023 Jan;33(1):1-6. doi: 10.1016/j.giec.2022.09.004. Epub 2022 Oct 23. PMID 36375876
- [Background] Maydeo A, Dhir V. Third-space endoscopy: stretching the limits. Gastrointest Endosc. 2017 Apr;85(4):728-729. doi: 10.1016/j.gie.2016.12.002. No abstract available. PMID 28317688
- [Background] Karanfilian B, Kahaleh M. New Applications for Submucosal Tunneling in Third Space Endoscopy: A Comprehensive Review. J Clin Gastroenterol. 2022 Jul 1;56(6):465-477. doi: 10.1097/MCG.0000000000001694. Epub 2022 Apr 1. PMID 35357336
- [Background] Bapaye A, Korrapati SK, Dharamsi S, Dubale N. Third Space Endoscopy: Lessons Learnt From a Decade of Submucosal Endoscopy. J Clin Gastroenterol. 2020 Feb;54(2):114-129. doi: 10.1097/MCG.0000000000001296. PMID 31851106
- [Background] Baars JE, Stoklosa T, Kaffes AJ, Saxena P. Maintaining hemostasis during third-space endoscopy. VideoGIE. 2018 Aug 8;3(10):304-305. doi: 10.1016/j.vgie.2018.07.004. eCollection 2018 Oct. No abstract available. PMID 30276349
- [Background] Li AA, Zhou MJ, Hwang JH. Understanding the Principles of Electrosurgery for Endoscopic Surgery and Third Space Endoscopy. Gastrointest Endosc Clin N Am. 2023 Jan;33(1):29-40. doi: 10.1016/j.giec.2022.07.001. PMID 36375884
- [Background] Akintoye E, Kumar N, Obaitan I, Alayo QA, Thompson CC. Peroral endoscopic myotomy: a meta-analysis. Endoscopy. 2016 Dec;48(12):1059-1068. doi: 10.1055/s-0042-114426. Epub 2016 Sep 12. PMID 27617421
- [Background] Stavropoulos SN, Modayil RJ, Friedel D, Savides T. The International Per Oral Endoscopic Myotomy Survey (IPOEMS): a snapshot of the global POEM experience. Surg Endosc. 2013 Sep;27(9):3322-38. doi: 10.1007/s00464-013-2913-8. Epub 2013 Apr 3. PMID 23549760
- [Background] Horikawa Y, Toyonaga T, Mizutamari H, Mimori N, Kato Y, Fushimi S, Okubo S. Feasibility of Knife-Coagulated Cut in Gastric Endoscopic Submucosal Dissection: A Case-Control Study. Digestion. 2016;94(4):192-198. doi: 10.1159/000450994. Epub 2016 Dec 9. PMID 27931026